CLINICAL TRIAL: NCT02254031
Title: An Open Phase I Dose Escalation Study of Bivatuzumab Mertansine Administered Intravenously Once Per Week for Three Weeks in Female Patients With CD44v6 Positive Recurrent or Metastatic Breast Cancer With Repeated Administration Courses in Patients With Clinical Benefit
Brief Title: Dose Escalation of Bivatuzumab Mertansine in Female Patients With CD44v6 Positive Recurrent or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1191.3
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — bivatuzumab mertansine

ARMS (1):
- bivatuzumab mertansine (Experimental): dose escalation
  Interventions: Drug: bivatuzumab mertansine

INTERVENTIONS:
Drug: bivatuzumab mertansine

SUMMARY:
maximum tolerated dose (MTD), safety, pharmacokinetics, efficacy of bivatuzumab mertansine

ELIGIBILITY:
Inclusion Criteria:

1. female patients aged 18 years or older
2. patients with breast cancer positive for CD44v6 in at least 50 % of the tumour cells
3. patients with local and / or regional recurrent disease or distant metastases who are refractory to anthracyclines and / or taxanes (unless contraindications to taxanes and / or anthracyclines) or not amenable to established treatments
4. measurable tumour deposits by one or more radiological techniques (MRI, CT)
5. life expectancy of at least 6 months
6. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
7. patients must have given written informed consent (which must be consistent with International Conference of Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation)

Exclusion Criteria:

1. hypersensitivity to humanised or murine antibodies, immunoconjugates or the excipients of the trial drugs
2. known secondary malignancy requiring therapy
3. active infectious disease
4. brain metastases requiring therapy
5. neuropathy grade 2 or above
6. absolute neutrophil count less than 1,500/mm3
7. platelet count less than 100,000/mm3
8. bilirubin greater than 1.5 mg/dl (> 26 μmol/L, système internationale (SI) unit equivalent)
9. aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 3 times the upper limit of normal
10. serum creatinine greater than 1.5 mg/dl (> 132 μmol/L, SI unit equivalent)
11. concomitant non-oncological diseases which are considered relevant for the evaluation of the safety of the trial drug
12. chemo- or immunotherapy within the past four weeks prior to treatment with the trial drug or during the trial (except for present trial drug)
13. radiotherapy to breast and thorax region within the past four weeks prior to treatment with the trial drug or during the trial
14. women who are sexually active and unwilling to use a medically acceptable method of contraception
15. pregnancy or lactation
16. treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
17. patients unable to comply with the protocol

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2003-07-01 (Actual); Primary Completion 2005-01-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | up to 6 months

SECONDARY OUTCOMES:
Incidence of adverse events | up to 14 days after last drug administration
  graded according to common toxicity criteria (CTC)
Number of patients with clinically significant findings in laboratory examinations | up to 14 days after last drug administration
Number of patients with clinically significant findings in vital signs | up to 14 days after last drug administration
Number of patients with development of Human Anti-Human Antibody (HAHA) | up to 14 days after last drug administration
Area under the serum concentration time curve from time zero to time point 168 hours (AUC0-168) | up to 168 hours
Area under the serum concentration time curve from time zero to the time of the last quantifiable drug concentration (AUC0-tz) | up to 14 days after last drug administration
Area under the serum concentration time curve from time point zero to infinity (AUC0-∞) | up to 14 days after last drug administration
Maximum serum concentration (Cmax) | up to 14 days after last drug administration
Time to reach maximum serum concentration (tmax) | up to 14 days after last drug administration
Terminal elimination half-life (t1/2) | up to 14 days after last drug administration
Mean residence time (MRT) | up to 14 days after last drug administration
Total body clearance (CL) | up to 14 days after last drug administration
Volume of distribution at steady state (Vss) | up to 14 days after last drug administration
Volume of distribution during the terminal elimination phase (Vz) | up to 14 days after last drug administration
Trough concentration at steady state (Cpre,ss) | up to 7 days after drug administration
Minimum serum concentration during the dosing interval τ at steady state (Cmin,ss) | up to 7 days after drug administration
Linearity index (LI) | up to 14 days after last drug administration
Accumulation factor (RA) | up to 14 days after last drug administration
Tumor response | up to 14 days after last drug administration
  according to response evaluation criteria in solid tumours (RECIST)

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency